CLINICAL TRIAL: NCT02994108
Title: Using Text Messaging to Increase HPV Vaccination Among Young Sexual Minority Men
Brief Title: txt2protect: Using Text Messaging to Increase HPV Vaccination Among Young Sexual Minority Men
Acronym: t2p
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary Gerend, Associate Professor, Behavioral Sciences and Social Medicine, College of Medicine, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21CA208329-01 (NIH); 1R21CA208329-01 (NIH)
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Human Papillomavirus
Keywords: Human Papillomavirus; Men Who Have Sex with Men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- txt2protect (Experimental): Content was delivered in 2 phases over 36 weeks. During Phase 1 (weeks 1-3), participants received 10-12 messages daily. During Phase 2 (weeks 4-36), message frequency decreased to monthly messages. Phase 1 content was presented in 3 modules. Module 1 addressed information about HPV infection and HPV vaccination. Module 2 addressed motivation to receive HPV vaccine. Module 3 addressed behavioral skills and self-efficacy for initiating and completing the 3-dose series (e.g., talking with their doctor about the vaccine). Phase 2 "booster" messages largely reinforced Phase 1 content to foster continued engagement with the program.
  txt2protect: Text messages sharing HIV/STI prevention information with a focus on HPV infection and vaccination.
  Interventions: Behavioral: txt2protect
- Sexual Health Control (Active Comparator): Content was delivered in 2 phases over 36 weeks. During Phase 1 (weeks 1-3), participants received 10-12 messages daily. During Phase 2 (weeks 4-36), message frequency decreased to monthly messages. Phase 1 content was presented in 3 modules; however, unlike the treatment group, content was topic-based rather than theory-based and focused on general sexual health. Module 1 addressed basic facts about HIV and sexually transmitted infections (STI), including HPV. Module 2 addressed HIV/STI prevention (e.g., condom use, PrEP) and will included basic facts about HPV vaccination currently available online. Module 3 addressed tips for healthy relationships. Phase 2 "booster" messages largely reinforced Phase 1 content to foster continued engagement with the program.
  Sexual Health Control: Text messages sharing HIV/STI prevention and healthy relationship building information, including information about HPV infection and vaccination.
  Interventions: Behavioral: Sexual Health Control

INTERVENTIONS:
Behavioral: txt2protect — Text messages sharing HIV/STI prevention information with a focus on HPV infection and vaccination.
  Other Names: t2p
  Arms: txt2protect
Behavioral: Sexual Health Control — Text messages sharing HIV/STI prevention and healthy relationship building information, including information about HPV infection and vaccination.
  Arms: Sexual Health Control

SUMMARY:
Human Papillomavirus (HPV) is a common sexually transmitted infection that can cause cancer (anal, penile, oropharyngeal) and genital warts in men. Due to their sexual practices (e.g., receptive anal intercourse), men who have sex with men (MSM) are at particularly high risk for HPV infection and are disproportionately affected by HPV-related cancers. A safe and effective vaccine is available to prevent HPV infection, yet HPV vaccination rates in the U.S. have been low, particularly among males. To remedy this gap, the goal of this study is to develop and pilot test a text messaging intervention to increase HPV vaccination in young MSM.

The study has two specific aims:

1. Develop, iteratively refine, and pre-test messages using a formative research procedure for designing targeted health interventions. The procedure consists of the following steps: 1) conduct online focus groups, an online survey, and in-depth interviews to inform message content, 2) draft initial messages based on focus group findings and pilot data, 3) refine message content and assess acceptability using content advisory teams, 4) conduct internal alpha testing to ensure software functionality, and 5) beta test the protocol.
2. Test the feasibility, acceptability, and preliminary efficacy of the txt2protect (t2p) text messaging intervention in a pilot randomized controlled trial (RCT). To achieve this aim, 460 unvaccinated MSM (ages 18-25) who live in the Chicago metro area will be randomly assigned to the treatment (t2p) or control condition. The treatment condition will receive a culturally appropriate text messaging-based HPV vaccination intervention based on the Information, Motivation, and Behavioral Skills model, whereas the control condition will receive a text messaging-based sexual health intervention that includes basic facts about HPV vaccination readily accessible online.

Primary outcome measures include intervention feasibility (e.g., retention in the trial), acceptability (satisfaction with the intervention), and preliminary efficacy as determined by initiation (receipt of the first dose) and completion of the 3-dose HPV vaccine series at the end of the 9-month trial.

The study team hypothesizes that participants in the t2p condition (vs. control) will report greater acceptability of the intervention and will be significantly more likely to initiate and complete the 3-dose HPV vaccine series by the end of the trial.

ELIGIBILITY:
Inclusion Criteria

Participants must:

1. Be male (sex at birth and gender identity)
2. Self-identify as gay, bisexual, or queer; ever had sex with a man; or be physically attracted to men
3. Be English speaking
4. Live in the Chicago metro area
5. Be the exclusive owner of a cell phone
6. Have used text messaging for at least 6 months
7. Plan to have the same cell phone number for the next 9 months
8. Be enrolled in an unlimited text messaging plan

Exclusion Criteria

* Participants must not have been previously vaccinated for HPV.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gerend, PhD, Principal Investigator — Florida State University; Brian Mustanski, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI agrees to develop a de-identified database, codebook, and mechanism by which IPD could be shared with other investigators upon approval of the PI. Data will be available for request approximately 6 months after completion of the project. Interested investigators will be asked to complete a standardized request form stating the specific aims of the analysis, the analytic plans, resources the requestors have to carry out the project, the proposed timeline, and distribution goals (manuscripts and/or grant application). The PI will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to undertake the request, how data will be protected/managed, and whether there are sufficient resources to honor the request. If any of these issues are problematic, the PI will attempt to negotiate a fair resolution with the interested parties and/or with NIH program staff.

REFERENCES:
- [Derived] Gerend MA, Madkins K, Crosby S, Korpak AK, Phillips GL, Bass M, Houlberg M, Mustanski B. Evaluation of a Text Messaging-Based Human Papillomavirus Vaccination Intervention for Young Sexual Minority Men: Results from a Pilot Randomized Controlled Trial. Ann Behav Med. 2021 Apr 7;55(4):321-332. doi: 10.1093/abm/kaaa056. PMID 32914838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment took place from January through early September 2018 in the Chicago area.
Pre-assignment Details: Although 155 participants completed the baseline survey, only 150 of them were randomized. A double screening protocol was used to ensure participants who had already been vaccinated were not accidentally enrolled. Five participants reported receiving a dose of HPV vaccine on baseline so they were no longer eligible for the RCT.
Period: Intervention Messages
Arm/Group | txt2protect | Sexual Health Control
Started | 74 | 76
Completed | 72 | 76
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Phase 1 Assessment
Arm/Group | txt2protect | Sexual Health Control
Started (Enrolled participants were allowed to complete follow-up even if they did not receive all messages.) | 72 | 76
Completed | 67 | 73
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3
Period: Phase 2 Assessment
Arm/Group | txt2protect | Sexual Health Control
Started (Enrolled participants were allowed to complete follow-up even if they did not receive all messages.) | 72 | 76
Completed | 63 | 69
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 8 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sexual Health Control: Content was delivered in 2 phases over 36 weeks. During Phase 1 (weeks 1-3), participants received 10-12 messages daily. During Phase 2 (weeks 4-36), message frequency decreased to monthly messages. Phase 1 content was presented in 3 modules; however, unlike the treatment group, content was topic-based rather than theory-based and focused on general sexual health. Module 1 addressed basic facts about HIV and sexually transmitted infections (STI), including HPV. Module 2 addressed HIV/STI prevention (e.g., condom use, PrEP) and will included basic facts about HPV vaccination currently available online. Module 3 addressed tips for healthy relationships. Phase 2 "booster" messages largely reinforced Phase 1 content to foster continued engagement with the program.
  Sexual Health Knowledge Control: Text messages sharing HIV/STI prevention and healthy relationship building information, including information about HPV infection and vaccination.
- Total: Total of all reporting groups
Arm/Group | txt2protect | Sexual Health Control | Total
Number analyzed (Participants) | 72 | 76 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 76 | 148
  >=65 years | 0 | 0 | 0
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 22.78 (2.03) | 23.06 (2.39) | 22.92 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 72 | 76 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 20 | 47
  Not Hispanic or Latino | 45 | 56 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 18 | 31
  White | 42 | 38 | 80
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 9 | 7 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 76 | 148
Sexual Orientation [Count of Participants; unit: Participants]
  Gay | 53 | 57 | 110
  Bisexual | 17 | 15 | 32
  Other (e.g., queer, pansexual) | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Intervention feasibility will be evaluated by retention in the RCT. The retention rate will be computed at the end of the 9-month trial by dividing the total number of participants who completed the trial (i.e., completed the 9-month assessment) by the total number of participants who were randomized to the treatment or control condition at the beginning of the trial. An 80% 9-month retention rate will be used to indicate a feasible intervention.
Time Frame: 9 Month
Population: A total of 150 participants were randomized. Three participants, all of whom were in the txt2protect arm, withdrew from the study. One of the three participants who withdrew provided permission to use include his data up until his withdrawal in month 3 and thus this participant was included in the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 72 | 76
Participants | 63 | 69
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .601, Chi-squared; Chi-Square = 0.415

2. Primary Outcome: Intervention Acceptability for Phase 1
Description: Intervention acceptability for the first 3 weeks of the intervention (Phase 1) will be assessed at the 3-week assessment. The scale includes both open-ended ("What did you like about the program? What could be improved?") and 12 closed-ended questions (e.g., "I would recommend a program like this to my friends" 1=strongly disagree to 5=strongly agree). Closed-ended items were combined to compute an average score (minimum value = 1; maximum value = 5). Higher scores indicate greater satisfaction with the program. An average score ≥4 will be used to indicate an acceptable intervention.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.25 (0.44) | 4.16 (0.49)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .249, t-test, 2 sided; Mean Difference (Final Values) = -0.09

3. Primary Outcome: Intervention Acceptability for Full Intervention
Description: Intervention acceptability for the full intervention will be assessed at the end the 9-month trial. The scale includes both open-ended ("What did you like about the program? What could be improved?") and 11 closed-ended questions (e.g., "I would recommend a program like this to my friends" 1=strongly disagree to 5=strongly agree). Closed-ended items will be combined to compute an average score (minimum value = 1; maximum value = 5). Higher scores indicate greater satisfaction with the program. An average score ≥4 will be used to indicate an acceptable intervention.
Time Frame: 9 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 63 | 69
score on a scale | 4.22 (0.51) | 4.18 (0.50)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .675, t-test, 2 sided; Mean Difference (Final Values) = -.04

4. Primary Outcome: Number of Participants Who Initiated the HPV Vaccine Series
Description: A final confirmatory assessment of HPV vaccination status will be conducted at the 9-month follow-up. Participants will be asked whether they received any doses of HPV vaccine (yes/no) since baseline and if yes, the number of doses and received. Vaccination status will be confirmed by consulting the Illinois Comprehensive Automated Immunization Registry (I-CARE). HPV vaccine initiation was defined as receipt of one or more doses of HPV vaccine by the end of the 9-month trial.
Time Frame: 9 Month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 72 | 76
Participants | 14 | 5
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .025, Regression, Logistic; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.17 to 10.08]

5. Primary Outcome: Number of Participants Who Completed the HPV Vaccine Series
Description: A final confirmatory assessment of HPV vaccination status will be conducted at the 9-month follow-up. Participants will be asked whether they received any doses of HPV vaccine (yes/no) since baseline and if yes, the number of doses received. Vaccination status will be confirmed by consulting the Illinois Comprehensive Automated Immunization Registry (I-CARE). HPV vaccine completion was defined as receipt of three doses of HPV vaccine by the end of the 9-month trial.
Time Frame: 9 Month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 72 | 76
Participants | 2 | 1
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .923, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.08 to 16.95]

6. Secondary Outcome: Information: HPV-related Knowledge
Description: Assessed with two questions (e.g., "HPV can cause anal cancer.") interspersed among other true/false questions assessing HIV/STI knowledge. Participants received one point for each correct response and zero points for incorrect and "don't know" responses. Points were summed to create a composite score that ranged from 0 to 2.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 1.11 (0.40) | 1.00 (0.50)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .174, t-test, 2 sided; Mean Difference (Final Values) = -0.11

7. Secondary Outcome: Motivation: Attitudes
Description: Assessed with one item: "My attitude toward getting vaccinated for HPV in the next 9 months is..." 1 = very negative to 5 = very positive.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.51 (0.61) | 4.11 (0.87)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .002, t-test, 2 sided; Mean Difference (Final Values) = -0.40

8. Secondary Outcome: Motivation: Subjective Norms
Description: Assessed with one item: "People who are important to me would want me to get vaccinated for HPV in the next 9 months." 1 = strongly disagree to 5 = strongly agree.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.10 (0.78) | 4.11 (0.94)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .964, t-test, 2 sided; Mean Difference (Final Values) = 0.01

9. Secondary Outcome: Motivation: Perceived Susceptibility
Description: Assessed with four items (e.g., "If you don't get the HPV vaccine, what do you think are the chances that you will get HPV?" 1 = very unlikely to 5 = very likely).
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 3.12 (1.00) | 2.78 (1.04)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .053, t-test, 2 sided; Mean Difference (Final Values) = -0.34

10. Secondary Outcome: Motivation: Perceived Severity
Description: Assessed with four items (e.g., "How serious would each of the following be for you: If you developed warts on your penis or scrotum?" 1 = not at all serious to 5 = very serious).
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.56 (0.49) | 4.66 (0.44)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .183, t-test, 2 sided; Mean Difference (Final Values) = 0.10

11. Secondary Outcome: Motivation: Anticipated Regret
Description: Assessed with two items (e.g., "How much regret would you feel if you decided not to get the HPV vaccine and later developed genital or anal warts?" 1 = none to 5 = quite a lot).
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.76 (0.60) | 4.50 (0.99)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .064, t-test, 2 sided; Mean Difference (Final Values) = -0.26

12. Secondary Outcome: Behavioral Skills: Perceived Behavioral Control
Description: Assessed with one item: "To what extent is whether or not you get vaccinated for HPV in the next 9 months under your control?" 1 = not at all to 5 = completely.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.42 (0.68) | 4.19 (1.07)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .147, t-test, 2 sided; Mean Difference (Final Values) = -0.22

13. Secondary Outcome: Behavioral Skills: Self-efficacy
Description: Assessed with one item: "Assuming you wanted to, how hard or easy would it be for you to get vaccinated for HPV in the next 9 months?" 1 = very hard to 5 = very easy.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 3.96 (0.98) | 3.67 (1.05)
Statistical Analysis 1: Comparison: txt2protect vs Sexual Health Control; Test type: Superiority; p = .096, t-test, 2 sided; Mean Difference (Final Values) = -0.29

14. Secondary Outcome: Behavioral Intentions
Description: Assessed with one item: "I intend to get vaccinated for HPV in the next 9 months." 1 = strongly disagree to 5 = strongly agree.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | txt2protect | Sexual Health Control
Number analyzed (Participants) | 67 | 73
score on a scale | 4.16 (0.86) | 3.75 (1.06)
Statistical Analysis 1: Comparison: txt2protect; Test type: Superiority; p = .013, t-test, 2 sided; Mean Difference (Final Values) = -0.41

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | txt2protect | Sexual Health Control
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/76
Other Adverse Events (participants affected / at risk) | 0/72 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02994108/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02994108/Prot_SAP_001.pdf